CLINICAL TRIAL: NCT03406884
Title: Autologous Cardiac Stem Cell Injection in Patients With Hypoplastic Left Heart Syndrome: An Open Label Pilot Study.
Brief Title: The CHILD Trial: Hypoplastic Left Heart Syndrome Study.
Acronym: CHILD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190743
Record Dates: First submitted 2017-12-20; First posted 2018-01-23 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: stem cells; pediatric
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Intervention Model Description: The first 10 participants will be enrolled in Group A to assess safety and feasibility. An additional 22 participants will be enrolled in Group B and will be randomized to either the Treatment or Control Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open label C-kit+ cells Group A (Experimental): Group A is an open-label treatment group determining safety and feasibility. Participants enrolled in this group will be receiving previously harvested c-kit+ cells during their Stage II BDCPA operation. Harvested c-kit+ cells will be injected into the right ventricle directly intramyocardially.
  Interventions: Biological: c-kit+ cells
- C-kit+ cells Group B (Active Comparator): Participants randomized to Group B Treatment Group will receive previously harvested c-kit+ cells during their Stage II BDCPA operation. Harvested c-kit+ cells will be injected into the right ventricle directly intramyocardially.
  Interventions: Biological: c-kit+ cells
- No Intervention Group (No Intervention): Participants randomized to Group B Control Group will receive only their standard of care (SOC) Stage II BDCPA operation without the injection of harvested c-kit+ cells.

INTERVENTIONS:
Biological: c-kit+ cells — The autologous c-kit+ cells will be harvested from participant's right atrial tissue obtained from participant's SOC Norwood Operation. The harvested c-kit+ cells containing up to a total of 12,500 cells/kg will be delivered through 6-10 intramyocardial injections of approximately 100uL per injection for a total volume of approximately 0.6 mL.
  Other Names: Autologous c-kit-positive cells (c-kit+ cells)
  Arms: C-kit+ cells Group B; Open label C-kit+ cells Group A

SUMMARY:
The objectives of this pilot study are to evaluate the feasibility and safety of intramyocardial injection of autologous c-kit+ cells during the Stage II Bidirectional Cavopulmonary Anastomosis (BDCPA) operation and to observe effects on clinical outcome including right ventricular myocardial function, severity of tricuspid regurgitation, incidence of serious adverse events, re-hospitalizations, changes in health status, the need for transplantation, or mortality.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study, subjects must meet all of the inclusion criteria:

  1. Subjects with hypoplastic left heart syndrome (HLHS) (all types) requiring Stage I Norwood operation.

     Exclusion Criteria:
* Candidates will be excluded from the study if any of the following conditions are met:

  1. Subjects undergoing the Stage I Norwood operation who do not have HLHS.
  2. Subjects requiring mechanical circulatory support immediately prior to Stage II BDCPA operation (within 5 days).
  3. Parent or guardian unwilling or unable to comply with necessary follow-up(s).
  4. Mother is serum positive for HIV 1/2, hepatitis B surface antigen or viremic hepatitis C and Treponema pallidum.
  5. Subjects who are unsuitable for inclusion in the study in the opinion of the investigator(s).

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University; Kristopher Deatrick, MD, Principal Investigator — University of Maryland; Richard Ohye, MD, Principal Investigator — Michigan Medicine Congenital Heart Center/C.S. Mott Children's Hospital
Locations (4):
- United States (4):
  - Emory University Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Maryland - Division of Cardiac Surgery, Baltimore, Maryland
  - Michigan Medicine Congenital Heart Center/C.S. Mott Children's Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaushal S, Hare JM, Mahle WT, Khan A, Ohye RG, Slesnick TC, Chai PJ, Shashidharan S, Robinson JD, Jone PN, Doman T, Si MS, Lu JC, Bacallao K, Nettina AE, Lamazares R, Saltzman RG, Simpson LM, Li R, Bettencourt JE, Mansoor K, Davis BR, Deatrick KB, Yang J, Mishra R, Everett AD, Lai D, Davis ME. Phase I Randomized Study of Cardiac Stem Cells in Patients With Hypoplastic Left Heart Syndrome: The CHILD Trial. JACC Heart Fail. 2026 Jan;14(1):102723. doi: 10.1016/j.jchf.2025.102723. Epub 2025 Nov 19. PMID 41258851
- [Derived] Kaushal S, Hare JM, Shah AM, Pietris NP, Bettencourt JL, Piller LB, Khan A, Snyder A, Boyd RM, Abdullah M, Mishra R, Sharma S, Slesnick TC, Si MS, Chai PJ, Davis BR, Lai D, Davis ME, Mahle WT. Autologous Cardiac Stem Cell Injection in Patients with Hypoplastic Left Heart Syndrome (CHILD Study). Pediatr Cardiol. 2022 Oct;43(7):1481-1493. doi: 10.1007/s00246-022-02872-6. Epub 2022 Apr 8. PMID 35394149
- [Derived] Ali MK, Ichimura K, Spiekerkoetter E. Promising therapeutic approaches in pulmonary arterial hypertension. Curr Opin Pharmacol. 2021 Aug;59:127-139. doi: 10.1016/j.coph.2021.05.003. Epub 2021 Jun 30. PMID 34217109
- See also: Interdisciplinary stem cell institute at the University of Miami website — http://ISCI.MED.MIAMI.EDU

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label C-kit+ Cells Group A: Group A is an open-label treatment group determining safety and feasibility. Participants enrolled in this group will be receiving previously harvested c-kit+ cells during their Stage II Bidirectional Cavopulmonary Anastomosis (BDCPA) operation. Harvested c-kit+ cells will be injected into the right ventricle directly intramyocardially.
  c-kit+ cells: The autologous c-kit+ cells will be harvested from participant's right atrial tissue obtained from participant's SOC Norwood Operation. The harvested c-kit+ cells containing up to a total of 12,500 cells/kg will be delivered through 6-10 intramyocardial injections of approximately 100 microliters per injection for a total volume of approximately 0.6 mL.
Period: Overall Study
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Started | 9 | 8 | 8
Completed | 9 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at BDCPA operation
  Months | 4.18 (0.57) | 4.66 (0.85) | 4.7 (0.89) | 4.51 (0.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 8 | 5 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 8 | 6 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 5
  White | 3 | 6 | 7 | 16
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Incidence of Treatment Related Major Adverse Cardiac Events
Description: Safety will be reported as the number of incidence of treatment related major adverse cardiac events (MACE). MACE is defined as any of the following: greater than 30 seconds of sustained/symptomatic ventricular tachycardia requiring intervention, cardiogenic shock, unplanned cardiovascular operation due to injection site bleeding, need for new permanent pacemaker, stroke or embolic event to the brain determined by CT scan and death. MACE will be evaluated by the treating physician and assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Time Frame: 30 days
Measure: Number; unit: Events
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
Events | 1 | 0 | 6

2. Primary Outcome: Number of C-kit+ Products
Description: Feasibility will be reported as the number of c-kit+ products that can be manufactured and delivered to subjects
Time Frame: Day 1
Measure: Number; unit: Products
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
Products | 9 | 7 | 0

3. Primary Outcome: Number of Participants Completing Magnetic Resonance Imaging (MRI)
Description: Feasibility will be reported as the number of participants that complete the baseline, 6-months, and 12-months follow up MRI.
Time Frame: Baseline, 6 Months, 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
Participants
  Baseline | 9 | 7 | 7
  Month 6 | 6 | 6 | 5
  Month 12 | 6 | 6 | 2

4. Primary Outcome: Change in Right Ventricular Function (RVEF)
Description: Efficacy will be reported as the change in right ventricular function assessed as a percentage and will be measuring using serial echocardiograms and MRI scan.
Time Frame: Baseline, 6 Months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
percentage
  Baseline: number analyzed (Participants) | 9 | 7 | 7
  Baseline | 49.33 (4.44) | 55 (7.19) | 45.4 (10.25)
  Month 6: number analyzed (Participants) | 6 | 6 | 5
  Month 6 | 48 (3.63) | 50.83 (6.74) | 47 (6.86)
  Month 12: number analyzed (Participants) | 6 | 6 | 2
  Month 12 | 44.67 (8.36) | 49.83 (3.76) | 48.5 (3.54)

5. Primary Outcome: Change in Right Ventricular End-diastolic Volume (RVEDV)
Description: Efficacy will be reported as the change in right ventricular end-diastolic assessed in milliliters per square meter and will be measured using serial echocardiograms and MRI scan.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: milliliters per square meter
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
milliliters per square meter
  Baseline: number analyzed (Participants) | 9 | 7 | 7
  Baseline | 112.57 (20.75) | 119.1 (35.08) | 123.98 (18.92)
  Month 6: number analyzed (Participants) | 6 | 6 | 5
  Month 6 | 129.5 (44.21) | 123.08 (11.83) | 130.27 (37.08)
  Month 12: number analyzed (Participants) | 6 | 6 | 2
  Month 12 | 126.78 (23.55) | 113.8 (13.97) | 129 (18.1)

6. Primary Outcome: Change in Right Ventricular End-systolic Volume (RVESV)
Description: Efficacy will be reported as the change in right ventricular end-systolic volume assessed in milliliters per square meter and will be measured using serial echocardiograms and MRI scan.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: milliliters per square meter
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
milliliters per square meter
  Baseline: number analyzed (Participants) | 9 | 7 | 7
  Baseline | 57.43 (13.22) | 55.53 (23.87) | 68.66 (22.04)
  Month 6: number analyzed (Participants) | 6 | 6 | 5
  Month 6 | 68.38 (26.43) | 55.17 (21.36) | 70.66 (28.95)
  Month 12: number analyzed (Participants) | 6 | 5 | 2
  Month 12 | 71.7 (21.64) | 56.66 (5.43) | 68.05 (12.8)

7. Primary Outcome: Change in Tricuspid Regurgitation
Description: Efficacy will be reported as the change tricuspid regurgitation assessed as a percentage and will be measured using serial echocardiograms and MRI scan.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
percentage
  Baseline: number analyzed (Participants) | 6 | 5 | 4
  Baseline | 8.28 (5.21) | 5 (0) | 5 (0)
  Month 6: number analyzed (Participants) | 3 | 4 | 4
  Month 6 | 35.07 (27.81) | 9.23 (6.03) | 15.35 (16.95)
  Month 12: number analyzed (Participants) | 3 | 5 | 2
  Month 12 | 21.93 (6.03) | 14.72 (7.27) | 7.75 (3.75)

8. Secondary Outcome: Number of Incidence of Serious Adverse Events
Description: Incidence of the following after the BDCPA / GLENN Procedure including: All-cause mortality; Cardiovascular mortality; Need for transplantation; Hospitalization for heart failure; Cardiovascular morbidity, including stroke or heart failure or sustained/symptomatic arrhythmias.
Time Frame: Up to 12 months
Measure: Number; unit: Events
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
Events | 1 | 0 | 6

9. Secondary Outcome: Change in Somatic Growth Velocity - Length (cm)
Description: Changes in somatic growth velocity will be evaluated by length (cm) over 12 months post study product injection.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
centimeters
  Baseline: number analyzed (Participants) | 9 | 7 | 7
  Baseline | 60.33 (3.82) | 59.5 (3.28) | 60.07 (4.94)
  Month 6: number analyzed (Participants) | 9 | 7 | 7
  Month 6 | 69.72 (5.57) | 69.79 (4.18) | 70.8 (5.39)
  Month 12: number analyzed (Participants) | 9 | 7 | 6
  Month 12 | 76.98 (5.87) | 77.03 (3.7) | 79.63 (4.02)

10. Secondary Outcome: Change in Somatic Growth Velocity - Weight (kg)
Description: Changes in somatic growth velocity will be evaluated by weight (kg) over 12 months post study product injection.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
kilograms
  Baseline: number analyzed (Participants) | 9 | 7 | 7
  Baseline | 5.7 (0.66) | 5.6 (0.74) | 5.65 (0.69)
  Month 6: number analyzed (Participants) | 9 | 7 | 7
  Month 6 | 7.67 (0.84) | 8.39 (1.21) | 8.36 (0.65)
  Month 12: number analyzed (Participants) | 9 | 7 | 6
  Month 12 | 9.74 (1.65) | 10.45 (1.19) | 10.01 (0.68)

11. Secondary Outcome: Change in Somatic Growth Velocity - Head Circumference (cm)
Description: Changes in somatic growth velocity will be evaluated by head circumference (cm) over 12 months post study product injection.
Time Frame: Baseline, 6 months, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
centimeters
  Baseline: number analyzed (Participants) | 9 | 6 | 7
  Baseline | 38.51 (3.01) | 39.58 (2.69) | 38.33 (3.18)
  Month 6: number analyzed (Participants) | 7 | 4 | 6
  Month 6 | 45.04 (1.33) | 45.18 (1.62) | 45.42 (2.42)
  Month 12: number analyzed (Participants) | 6 | 6 | 5
  Month 12 | 47.88 (0.76) | 48.48 (1.57) | 46.92 (2.39)

12. Secondary Outcome: Change in Infant Toddler Quality of Life Survey (ITQOL) - Overall Health
Description: The Infant Toddler Quality of Life Survey (ITQOL) is a validated 47-item parent-reported questionnaire assessing multiple domains of child health, including overall health, physical abilities, growth and development, discomfort/pain, mood, and behavior. Domain scores are transformed to a 0-100 scale, where 0 reflects the poorest health-related quality of life and 100 reflects the best. Higher scores indicate better quality of life.
Time Frame: Baseline, 12 months
Population: sample size decreases due to attrition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
score on a scale
  Baseline: number analyzed (Participants) | 5 | 7 | 7
  Baseline | 86 (16.36) | 62.14 (24.64) | 77.86 (12.2)
  Month 12: number analyzed (Participants) | 5 | 7 | 6
  Month 12 | 88 (6.71) | 85.71 (13.36) | 72.5 (13.69)

13. Secondary Outcome: Incidence of Mortality or Need for Transplantation
Description: Incidence of mortality or need for transplantation after the Stage II BDCPA operation will be reported
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
Number analyzed (Participants) | 9 | 8 | 8
Participants | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Open Label C-kit+ Cells Group A | C-kit+ Cells Group B | No Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 1/8
Serious Adverse Events (participants affected / at risk) | 8/9 | 4/8 | 4/8
Other Adverse Events (participants affected / at risk) | 5/9 | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label C-kit+ Cells Group A (N=9) | C-kit+ Cells Group B (N=8) | No Intervention Group (N=8)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Crying (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aortic restenosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Infant irritability (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Collateral circulation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label C-kit+ Cells Group A (N=9) | C-kit+ Cells Group B (N=8) | No Intervention Group (N=8)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Device embolisation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Medication Error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery occlusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03406884/Prot_SAP_000.pdf